CLINICAL TRIAL: NCT06747624
Title: A Crossover Clinical Trial Investigating the Effects of Geranylgeraniol (GG) Supplementation on Testosterone Levels in Healthy Men and Women Over an 18-week Period
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Designs for Health (Industry)
Responsible Party: Principal Investigator, Michael Jurgelewicz, Director, Product Development, Research, and Clinical Support, Designs for Health
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AR - 30040
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Wellness; Health
Keywords: Geranylgeraniol; GG
MeSH Terms: interventions — geranylgeraniol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Geranylgeraniol 300 mg (Experimental)
  Interventions: Dietary Supplement: Geranylgeraniol 300 mg
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Geranylgeraniol 300 mg — 300 mg of trans-geranylgeraniol (GG)
  Arms: Geranylgeraniol 300 mg
Dietary Supplement: Placebo — 300 mg medium chain triglycerides
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to investigate the effects of geranylgeraniol (GG) supplementation on testosterone levels in middle-aged (40 to 65 years) healthy men and women.

The research team hypothesizes that geranylgeraniol (GG) supplementation will enhance testosterone levels and improve self-reported health outcomes in a healthy population.

DETAILED DESCRIPTION:
The proposed study is an 18-week crossover, placebo-controlled pilot study of GG supplementation or placebo. All study outcomes will be measured at baseline (the beginning of the first week) and at the conclusion of the first 8-week period. This will be followed by a 2-week washout period; study procedures will be repeated with the second intervention for an additional 8 weeks. Outcomes will be assessed at the beginning of this period, and the end, in the same manner as for the first 8-week block.

All participants will receive a placebo (300 mg medium chain triglycerides/daily) or gernaylgeraniol supplementation (300 mg GG/daily). Subjects will be required to fast for 8 hours with no alcohol consumption before their blood draw. Baseline blood samples will be drawn before administering one of two treatments with subsequent blood samples to be drawn in the morning (between 7 am and 8 am) at 8, 10, and 18 weeks. Each participant will take the assigned intervention daily with breakfast for the following 8 weeks. After a 14-day washout period, this process will be repeated for the remaining treatment. Self-reported height and weight will be obtained to calculate body mass index (BMI). Questionnaires on overall health (SF-36) and sexual health [PROMIS Sexual Function and Satisfaction (SexFS) v2.0 Brief Profile (Male/Female)] will be assessed at baseline, 8, 10, and 18 weeks. All laboratory testing will occur at a LabCorp patient service center. The serum samples will be analyzed for Free and Total Testosterone using liquid chromatography with tandem mass spectrometry (LC-MS-MS). LabCorp test code: 070195; Serum Sex Hormone-Binding Globulin (SHBG) will be analyzed using Electrochemiluminescence immunoassay (ECLIA). LabCorp test code: 082016. Coenzyme Q10, Total (CoQ10). LabCorp test code: 120251.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 40 to 65 years of age.
2. Individuals with no significant history of inflammatory bowel disease (i.e. ulcerative colitis, Crohn's, Celiac, etc.), ulcers, liver and/or kidney disease or other any acute or chronic dis-ease.
3. Ability to read and speak English
4. Subject's agreement to voluntarily participate in the study
5. Negative pregnancy test confirmed with serum HCG on initial baseline testing and baseline testing at the start of the crossover (at 10 weeks)

Exclusion Criteria:

1. Males and females under 40 or over 65 years of age
2. Previous (in the past 60 days) or current hormone replacement therapy
3. Males and females with free testosterone levels over normal range
4. History of hysterectomy, oophorectomy, or orchiectomy
5. Current biotin supplementation >3 mg per day one week prior to the start of the study
6. Current or history of smoking
7. CoQ10/Ubiquinol supplementation within the past 2 weeks
8. Current use of hormone boosting supplements (i.e. fenugreek, shilajit, tongkat ali, ashwagandha) within the past 4 weeks
9. Current or previous use of medication - NSAIDS, statins, blood thinners, H2 blockers and PPI or blood sugar-lowering agents.
10. Diabetes
11. Cancer
12. Hemophilia
13. Disorders of heart, kidney, lung or liver function
14. Infectious diseases
15. Alcohol or drug abuse (>7 drinks per week for men and women)
16. Pregnancy, lactation, or individuals planning to become pregnant in the next 6 months
17. Failure to submit statement of consent
18. Participant in a clinical trial in the previous 30 days.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Serum Total Testosterone (LC/MS-MS) | Baseline, 8 weeks, 10 weeks, and 18 weeks
  Can aid in the diagnosis of androgen dysfunction in men and women and is more specific method of measuring testosterone concentrations. Units in ng/ml.
Serum Free Testosterone (Direct) | Baseline, 8 weeks, 10 weeks, and 18 weeks
  The concentration of unbound testosterone in serum. The majority of serum total testosterone is associated with sex hormone binding globulin (SHBG) and this fraction is tightly bound and bio-logically unavailable to its target tissues. The remaining bioavailable testosterone is mostly bound to albumin, with only a small fraction circulating in the free form. Free testosterone is the form of testosterone that can diffuse into the tissues and act on receptors and is considered the active fraction. Free testosterone assessment is recommended as a primary or secondary measure of androgen activity in men and women. Units in pg/ml.

SECONDARY OUTCOMES:
Serum Sex Hormone Binding Globulin (SHBG) | Baseline, 8 weeks, 10 weeks, and 18 weeks
  The blood transport protein for testosterone and estradiol. SHBG binds reversibly to sexual steroids and is an important indicator of an excessive/chronic androgenic action where androgen levels are normal, but where clinical symptoms would seem to indicate androgen in excess. SHBG is a useful supplementary parameter in the determination of androgen where a high concentration of free androgen (i.e., testosterone) is suspected. Reference ranges in men: 20-49 years: 16.5-55.9 nmol/L; >49 years: 19.3-76.4 nmol/L. Reference ranges in women: 20-49 years: 24.6-122.0 nmol/L; >49 years: 17.3-125.0 nmol/L.
Coenzyme Q10 (CoQ10) | Baseline, 8 weeks, 10 weeks, and 18 weeks
  CoQ10 is endogenously synthesized via the mevalonate pathway and some is obtained in the diet from meat products. It is also a powerful lipid-soluble antioxidant protecting cell membranes and lipoproteins. Reference range: 0.37-2.20 µg/mL.
SF-12- Health Survey | Baseline, 8 weeks, 10 weeks, and 18 weeks
  The SF-12 (Short Form Health Survey) is an indicator of overall health status across eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.
PROMIS- Sexual Health and Satisfaction | Baseline, 8 weeks, 10 weeks, and 18 weeks
  Sexual health [PROMIS Sexual Function and Satisfaction (SexFS) v2.0 Brief Profile (Male) and (Female)]. The SexFS assesses interest in sexual activity. These are domains relevant to healthy individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Designs for Health, Inc., Palm Coast, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes